CLINICAL TRIAL: NCT00401921
Title: A Randomized, Placebo-Controlled Study of the Effects of Minocycline on Cognitive Function After Carotid Endarterectomy
Brief Title: A Study of the Effects of Minocycline on Cognitive Function After Carotid Endarterectomy
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: PI moved to a new facility
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Joanne O'Hara, Sr. Project Manager, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2006-P-001225
Record Dates: First submitted 2006-11-17; First posted 2006-11-22 (Estimated); Last update posted 2017-07-14 (Actual); Status verified 2017-07

CONDITIONS: Carotid Stenosis
MeSH Terms: conditions — Carotid Stenosis | interventions — Minocycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Minocycline arm (Placebo Comparator): Minocycline 100mg/Placebo 0mg Minocycline 100mg, 1 capsule PO BID starting 36 hours prior to surgery. 2 capsules the morning of surgery
  Interventions: Drug: Minocycline
- Placebo arm (Placebo Comparator): Placebo 0mg, 1 capsule PO BID starting 36 hours prior to surgery. 2 capsules the morning of surgery.
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Minocycline — 100 mg, 1 capsule PO BID starting 36 hours prior to surgery. 2 capsules the morning of surgery
  Other Names: Minocycline 100mg/Placebo 0mg
  Arms: Minocycline arm
Drug: Placebo oral capsule — 1 capsule PO BID starting 36 hours prior to surgery. 2 capsules the morning of surgery.
  Arms: Placebo arm

SUMMARY:
The primary aim of this protocol is to investigate a possible new, neuroprotective treatment to prevent cognitive deficits that occur after carotid endarterectomy. We will investigate whether a widely used antibiotic agent - minocycline - that has shown neuroprotective effects in animal models of neurological diseases - can reduce the cognitive deficits associated with the surgical procedure of carotid endarterectomy (CEA). Because these cognitive deficits are believed to be a result of small strokes (due to emboli and/or hypoperfusion), this study will provide preliminary data on the use of this drug as a neuroprotective agent in stroke - a leading cause of disability.

(1) The first aim of this study is to examine whether 5 doses of minocycline administered 36 hrs before and 1 dose 12 hrs after the surgical procedure in patients undergoing CEA are effective to reduce the cognitive deficits associated with this procedure as compared with placebo.

a. The null hypothesis is that there is no difference in cognitive performance changes after CEA between the patients that receive placebo or minocycline.

DETAILED DESCRIPTION:
This protocol is a phase IIa study that will prospectively investigate whether minocycline (an antibiotic that showed neuroprotective effects in animal models) can decrease the cognitive deficits associated with carotid endarterectomy. This trial will be a randomized, parallel-group design, double-blind, placebo controlled clinical trial conducted at the Brigham and Women's Hospital.

The principal aim of this investigation is to study the effects of minocycline on cognitive performance after carotid endarterectomy. To measure cognitive function, we will perform a neuropsychological battery of tests (as detailed below). This battery of tests will be carried out by a blinded rater (a neurologist) and will be performed according to the following timetable:

Training session: before the baseline, patients will perform the tasks several times until they reach a stable plateau (defined as a variation of less than 10% in the last three trials) in order to eliminate the confounding effect of learning.

Baseline evaluation: the baseline evaluation will be performed in the day prior to the surgery.

Post-treatment evaluation: post-treatment evaluation will be performed 24 hours after the surgical procedure by the same blinded rater.

Neuropsychological battery of tests: we based our neuropsychological battery of tests on a similar study that evaluated the cognitive deficits associated with CEA and will consist of the following tests:

1. Trail making test - parts A and B (this test evaluates visual concept and visuo-motor track)
2. Controlled Oral Word Association (letters C, F and L) (this test evaluates verbal fluency)
3. The Boston Naming Test (naming of 60 pictures) (this test evaluates left hemisphere damage)
4. Digit Span Forward and Backward (this test evaluates working memory)
5. Stroop Task (this test evaluates selective attention and mental flexibility)
6. Mini-mental state examination (this test evaluates an adult patient's level of global cognitive functioning)

Blood sample analysis: As a secondary outcome, we will analyze subjects blood sample in respect to two particular substances: S100B and neuron specific enolase. The rationale for performing proteomic studies is that past research has shown that subtle cerebral injuries after carotid endarterectomy, even in the absence of stroke, might be associated with a significant increase in serum S100B (Connolly, 2001 - Neurosurgery, 2001 49 (5)) and also in traumatic brain injury (Cotena, 2006, J Neurosurg 2006 104 (6)). In addition, neuron specific enolase (NSE) also seems to be valuable to predict brain damage in patients with brain traumatic injury (Naeimi, 2006 - Brain Inj 2006 20(5)), thus showing that these two substances might be important biomarkers to be investigated in our study.

After eligibility screening (inclusion and exclusion criteria), consent form, medical history and physical exam participants will be randomized to the exposure - minocycline or placebo. The pills (minocycline and placebo) will have the same appearance and only one person will know whether the treatment is active or placebo.

Randomization:

Because our sample size will be relatively small, participants will be randomized to minocycline or placebo through a randomization stratification approach. This approach will ensure that both groups will have a similar distribution regarding baseline performance in the cognitive tests. Participants will be gathered into groups (strata) defined by their performance in the neuropsychological tasks (baseline). Participants within each stratum will be randomized to one of two treatment groups - minocycline and placebo - according to a block randomization of four and using a randomization list generated by a computer that will take into account the study entrance order. These groups are defined as follows:

Minocycline: we will use the dosage of minocycline that is currently used for clinical indications and also used in trials employing this drug as an anti-inflammatory agent. Minocycline will be administered in the period of 36 hrs before surgery (100 mg twice a day and 200 mg in the morning of the surgery - total of 5 doses) and 12 hrs after surgery (single dose of 100 mg).

The two doses of minocycline administered in the morning of the surgery will be taken with a small sip of water.

Placebo: placebo pill will have the same appearance as the real drug (minocycline) and will be administered using the same timetable as the active drug.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with carotid stenosis 60% or more with a clinical indication of CEA.
2. Patients that can perform the tests in English.
3. Women of childbearing age must be non-lactating and surgically sterile or using an effective method of birth control and have a negative pregnancy test (adequate birth control includes use of intra uterine device, or a barrier method, e.g. condom, diaphragm).
4. Ages Eligible for Study: 18 Years - 90 Years
5. Genders Eligible for Study: Both

Exclusion Criteria:

1. Known hypersensitivity to tetracyclines
2. Advanced cardiac, pulmonary or renal disease as assessed by the PCP of the patient.
3. Previous strokes with important clinical neurological deficits.
4. Pregnancy, breast-feeding or lactating
5. Baseline MMSE score less or equal to 20.
6. Female subjects on oral contraceptives.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-10; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Neuropsychological assessment | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Robert Friedlander, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States